CLINICAL TRIAL: NCT04337606
Title: Chidamide in Combination With Decitabine in Non-Hodgkin's Lymphoma Relapsed After Chimeric Antigen Receptor : An Open-label Phase I/II Trial
Brief Title: Chidamide in Combination With Decitabine in Non-Hodgkin's Lymphoma Relapsed After Chimeric Antigen Receptor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-046
Record Dates: First submitted 2020-04-04; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Decitabine; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chidamide in combination with decitabine (Experimental): chidamide 10mg/day, days 1-5, 20mg/day, day 8, 11,15, 18; decitabine 10 mg/day, days 1-5, every 3 weeks
  Interventions: Drug: Chidamide; Drug: Decitabine
- decitabine in combination with Camrelizumab (Experimental): decitabine 10 mg/day, days 1-5, every 3 weeks; camrelizumab 200mg d6
  Interventions: Drug: Decitabine; Drug: Camrelizumab

INTERVENTIONS:
Drug: Chidamide — Chidamide is a novel and orally active benzamide class of HDAC inhibitor that selectively inhibits activity of HDAC1, 2, 3 and 10, which can Induce tumor-cell apoptosis, suppress cell proliferation and enhance immune surveillance; Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1(DNMT1), which can increase tumor antigens and HLA expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function.
  Arms: chidamide in combination with decitabine
Drug: Decitabine — Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1(DNMT1), which can increase tumor antigens and HLA expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function.
Drug: Camrelizumab — Camrelizumab is a humanized anti-PD-1 monoclonal antibody.
  Arms: decitabine in combination with Camrelizumab

SUMMARY:
This is a Phase I/II clinical trial for patients with r/r Non-Hodgkin's Lymphoma relapsed after chimeric antigen receptor T cells infusion. The purpose is to evaluate the safety and efficacy of the treatment with chidamide in combination with decitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histological confirmation of Non-Hodgkin lymphoma (NHL) and relapsed after chimeric antigen receptor T cells infusion.
2. 18 to 65 years of age.
3. ECOG performance of less than 2.
4. Life expectancy of at least 3 months.
5. Subjects with lymphoma must have at least one measureable new lesion >1.5cm as defined by lymphoma response criteria.
6. Subjects must have relapsed after chimeric antigen receptor T cells infusion without any intervention treatment prior to Day 1.
7. Subjects must have adequate marrow, live, renal and heart functions.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in one month .
4. Prior organ allograft.
5. Women who are pregnant or breastfeeding.
6. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
7. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-04 (Estimated); Primary Completion 2024-04-04 (Estimated); Study Completion 2026-04-04 (Estimated)

PRIMARY OUTCOMES:
CR rate | 2 years
  CR rate assess by investigators per the 2014 Lugano classification rate of subjects achieved complete response in all evaluable subjects
Adverse events | 2 years
  Adverse events were defined according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China